CLINICAL TRIAL: NCT06428812
Title: Phd Student Msc Midwife
Brief Title: The Effect of Perineal Protective Package Application on Pelvic Floor in Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Öznur Hayat Öktem (Other)
Responsible Party: Sponsor-Investigator, Öznur Hayat Öktem, Phd student Msc midwife, Gulhane School of Medicine
Organization: Gulhane School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Hayatoktem02
Record Dates: First submitted 2024-05-15; First posted 2024-05-24 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Pregnancy; Labor; Pelvic Floor

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- perineal package application group (Experimental): This group includes those in the 2nd stage of labor upright position spontaneous pushing Hot application will be made
  Interventions: Other: Experimental: perineal package application group
- Routine hospital care (No Intervention): Routine hospital care

INTERVENTIONS:
Other: Experimental: perineal package application group — This group includes those in the 2nd stage of labor upright position spontaneous pushing Hot application will be made
  Arms: perineal package application group

SUMMARY:
This study aimed to evaluate the effect of perineal protection package application on labor outcomes, perineal integrity, postpartum urinary incontinence and pelvic floor muscle strength.In this study, a package including practices that have been proven to protect the perineum in labor was created and it was aimed to examine the effect of this perineal protection package; as a whole. The;perineal protective package; applications created by the researchers consisted of positioning on the gynecologic table (the back of the table was erected, the legs were removed from the hooks and placed on the sides of the table), open glottis pushing instead of closed glottis pushing, hot compress protection of the perineum instead of dry compress protection of the perineum, instead of lithotomy position in the second stage, which reduces the tension of the perineum and allows it to be observed and protected manually.

DETAILED DESCRIPTION:
The pelvic floor plays a critical and important role in maintaining healthy functions of the urinary, genital and gastrointestinal systems. When tissues in a region of the pelvic floor are damaged for any reason, pelvic floor dysfunction develops.

Pregnancy and childbirth are important risk factors for pelvic floor dysfunction. Hormonal and mechanical changes during pregnancy predispose to impaired pelvic floor function. During pregnancy, weight gain and increase in uterine weight increase intra-abdominal pressure. Therefore, ligaments and pelvic floor muscles are overstretched. He states that the main factor in pelvic floor dysfunction is vaginal delivery and that the passage of a particularly large fetal head through the birth canal is the trigger. During the passage and descent of the fetal head through the vaginal canal, the pelvic floor muscles can be overstretched, torn or damaged. Obstetric factors that cause pelvic floor damage include early or late age at first birth, high body mass index, large baby, length of the second stage of trauma (labor), forceps, vacuum, episiotomy and fundal compression.

Damage to the pelvic floor during labor has many short- and long-term effects on a woman's quality of life. These can be summarized as chronic perineal pain, pelvic organ prolapse, urinary and anal incontinence, fistula, sexual dysfunction, labor dissatisfaction, physical and psychological morbidities, and decreased quality of life. In addition, breastfeeding and mother-infant attachment problems may also occur due to perineal pain in the early postpartum period. Therefore, it is important to prevent pelvic floor damage in childbirth, which negatively affects physical, social and psychological well-being and leads to many short and long-term morbidities. The World Health Organization recommends the use of techniques such as hot compresses to reduce perineal damage and facilitate spontaneous delivery.

In the literature, there are many studies examining interventions to protect the pelvic floor in labor. Studies show that perineal massage, perineal warm application, birth positions, hand maneuvers, pushing techniques, and limited episiotomy reduce the incidence of perineal injury.

However, studies on these techniques and practices are generally studies investigating the effectiveness of a single method. In a recent qualitative study, midwives were asked to evaluate the effect of some protective practices called; perineal package; as a whole. However, in this study, midwives; own practices and opinions were evaluated, and their effects on the pelvic floor or labor were not examined. International organizations recommend the application of evidence-based, perineal, and pelvic floor supportive and protective methods to pregnant women in labor. However, the relationship between these practices and postpartum pelvic floor muscle strength and the presence of incontinence, which are indicators of pelvic floor damage, is unclear and studies to evaluate this relationship are limited.

The research will be conducted in 4 stages. In Phase 1, pregnant women who meet the inclusion criteria will be interviewed when they are admitted to the delivery room. In the first interview, the relevant sections of the data collection form will be filled out, pelvic floor muscle strength will be measured with a perineometer, and the IIQ-7 and UDI-6 scales will be filled out. Pregnant women with incontinence detected in these scales will be excluded. Then, pregnant women will be randomized using the true random number generation method on the random.org website and assigned to the study and control groups. Then, the delivery process of all pregnant women in the study and control groups will be monitored and recorded using the relevant section of the data collection form.

In phase 2, the perineal pain felt by pregnant women in both groups will be evaluated using VAS when the second stage of labor begins. The second stage of labor is the time from complete dilatation of the cervix until the fetal head is born. During this stage, the study group will receive a perineal protection package while the control group will receive routine care. Postpartum perineal pain, episiotomy length if episiotomy was applied and perineal length will be measured in both groups. The results of the trauma will be recorded in the labor follow-up form.

In the 3rd stage, pregnant women in both groups will be interviewed at the 1st hour postpartum and perineal pain will be evaluated with VAS.

In the 4th stage, the pregnant women in the study and control groups will be measured pelvic muscle strength with a perineometer, perineal length will be measured and recorded on the relevant form during routine hospital control at the 6th week postpartum. UDI-6 (urinary distress inventory) and IIQ-7 (incontinence impact questionnaire) will be completed.

ELIGIBILITY:
Inclusion Criteria:

* 18- 35 years old
* Primipar
* Singleton pregnancy in the vertex position between 38 and 42 weeks
* A reactive NST tracing
* Without a systemic disease (heart, HT, diabetes)
* No problem speaking and understanding Turkish
* Who agreed to participate in the study

Exclusion Criteria:

* Obese pregnant women
* Pregnant women who gained more than 25 kilograms during pregnancy
* Multiple pregnancies
* Pregnant women with a neurological disease affecting the pelvic floor
* Pregnant women who have undergone pelvic surgery
* Contraindications for normal delivery (placenta previa, anomalies of presentation, etc.)
* Estimated fetal weight of 4000 g or more
* Who wants to opt out of the study
* Pregnant women who are scheduled for cesarean section at any time of trauma

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2024-07-08 (Actual); Primary Completion 2025-03-11 (Actual); Study Completion 2025-03-11 (Actual)

PRIMARY OUTCOMES:
Perineal muscle strengt | On initial admission to the delivery room and after 6 weeks postpartum
  Perineal muscle strength will be measured in cmH2o with a perineometer.
Perineal Pain | 1st hour postpartum
  Perineal pain will be assessed by VAS at the beginning and end of the second stage of labor and at the end of the 1st hour postpartum.

SECONDARY OUTCOMES:
Episiotomy and laseration status | 1st hour postpartum
  Episypotomy will be measured in cm with a paper ruler according to the application status.
Urinary incontinence status | 6 weeks postpartum
  Urinary incontinence status will be measured with UDI-6 and IIQ-7.

CONTACTS AND LOCATIONS:
Overall Officials: Nazan KARAHAN, Associate professor, Study Director — Gulhane School of Medicine; MEHMET BÜLBÜL, Associate professor, Principal Investigator — Karabuk University
Locations (1):
- Karabuk Training and Research Hospital, obstetrics clinic, Karabük, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] undefined